CLINICAL TRIAL: NCT03308344
Title: Promoting Wellbeing in Military Spouses With Training
Brief Title: Mindfulness Training in Military Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Amishi Jha, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20120295
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into three groups: (i) a mindfulness training with spouse trainers (MT-ST, n = 60) that will receive the training from peers who underwent an extensive training practicum; (ii) a mindfulness training with mindfulness expert trainer group (MT-ME, n = 30) that will receive the training from a mindfulness expert trainer; and (ii) a wait-list control group (WLC, n = 30) that will be tested before and after a no-training interval and may receive MT at a later time after their second testing if they are interested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spouse Trainers (MT-ST) (Experimental): Participants will engage in a short-form mindfulness training delivered by their peers who underwent an extensive training practicum.
  Interventions: Behavioral: Mindfulness training
- Wait-list control (No Intervention): Participants will be tested before and after a no-training interval and may receive training at a later time.
- Mindfulness Expert (MT-ME) (Experimental): Participants will engage in a short-form mindfulness training delivered by an expert mindfulness trainer.
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — The present MT program includes topics related to mindfulness, emotion regulation, and connection. It will be delivered in short, weekly sessions.
  Arms: Mindfulness Expert (MT-ME); Spouse Trainers (MT-ST)

SUMMARY:
This project aims to contextualize the delivery of mindfulness training for military spouses and evaluate its effectiveness on measures of executive functions and psychological well-being.

DETAILED DESCRIPTION:
In addition to psychological and physical health challenges that military service members face, military deployment is known to have deleterious effects on the entire family unit. The January 2010 issue of the New England Journal of Medicine reported medical data from over 250,000 wives of deployed soldiers. These women suffered from clinically significant levels of anxiety, depression, sleep disturbances, and adjustment disorders. Thus, the psychological profile of military spouses sadly parallels that of the military servicemembers. Unfortunately, the effect of deployment on the psychological health in military spouses is largely unstudied, and very few resilience-building programs are available for military families.

Prior research showed that mindfulness training (MT), as a resilience-building program in civilian and military servicemembers, can effectively protect against degradation in of executive functions (i.e., attention, working memory) and benefit psychological well-being over high-demand intervals. While research evidence mounts that MT is beneficial for service members, there is almost no research examining the impact of MT on military spouses' cognitive functioning and psychological well-being.

The present study aims to investigate if MT may successfully benefit cognitive functioning and psychological well-being in military spouses.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Being in a relationship or married to U.S. Army active-duty member or veteran.

Exclusion Criteria:

* A non-controlled severe medical disease that might interfere with the performance in the study.
* Any other condition that the investigator might deem problematic for the inclusion of the volunteer in a training study of this nature.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Sustained Attention to Response Task (SART) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  SART is used to assess attentional performance and mind wandering. The task uses a continuous performance paradigm involving button presses to frequently presented non-targets (numbers 1, 2, 4, 5, 6, 7, 8, and 9) but requires the participants to withhold their motor response to the infrequent target (number 3). The subjective experience of mind wandering during SART is assessed through experience sampling probes randomly presented throughout the task.
Change in Working Memory task (WM) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  WMMW is used to assess working memory performance

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Scale (PANAS) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  PANAS assesses positive and negative affect. It consists of a list of descriptors of positive (e.g., 'interested', 'enthusiastic') and negative (e.g., 'irritable', 'upset') affects. Items are rated on a 5-point scale (1 = very slightly or not at all, 5 = extremely), according to how participants feel. The Positive Affect scale reflects the extent to which a person feels enthusiastic, active, and alert; the Negative Affect scale reflects unpleasant mood states, such as anger, disgust, and fear.
Change in Perceived Stress Scale (PSS) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  PSS assesses the degree to which situations in one's life are viewed as stressful within the past month. Individual items assess feelings of stress, nervousness, irritation at life's hassles, and perceptions of one's own coping and control over a situation.
Change in Self-Compassion Scale (SCQ) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  SCQ assesses self-compassion.
Change in Center for Epidemiological Studies Depression Scale (CES-D) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  This 20-item scale measures the major components of depressive symptomatology in the general population (i.e., nonpsychiatric persons older than 18).
Change in Anxiety Sensitivity Index (ASI) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  ASI assesses the construct of anxiety sensitivity.
Change in Perseverative Thoughts Questionnaire (PTQ) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  PTQ assesses stress due to reoccurring thoughts
Change in Marital Satisfaction | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  Marital Satisfaction questionnaire assesses the level of marital satisfaction.
Practice Logs | Participants will complete paper practice logs tracking their daily practice (i.e., minutes) from the beginning through the study completion, which is an average of 5 weeks after the beginning of the intervention.
  Practice logs will be used to keep track of participants' daily mindfulness practice.
Demographic Questions | Demographic questions will only be asked at the pre-intervention baseline (testing 1).
  General demographic questions will be asked to gather information about the participants, i.e. gender, age, partner ranking, partner deployment status etc.
Change in Cognitive Failures Questionnaire (CFQ) | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  CFQ assesses one's attention and awareness.
Feedback regarding the training | Feedback questions will be asked only at the second testing session (testing 2), which is an average of 5 weeks from the baseline.
  If participants were part of any of the training groups, they will be asked to provide feedback of the training.
Feedback regarding the testing | Feedback questions will be asked only at the second testing session (testing 2), which is an average of 5 weeks from the baseline.
  A 10-item questionnaire for participants to express their views and motivations about the tasks completed during the testing session.
General questions regarding life tendencies | Change from the pre-intervention baseline (testing 1) to post-intervention (testing 2), which is an average of 5 weeks from the baseline.
  General questions regarding life tendencies in a variety of situations during the past two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi Jha, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha AP, Morrison AB, Dainer-Best J, Parker S, Rostrup N, Stanley EA. Minds "at attention": mindfulness training curbs attentional lapses in military cohorts. PLoS One. 2015 Feb 11;10(2):e0116889. doi: 10.1371/journal.pone.0116889. eCollection 2015. PMID 25671579
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Mansfield AJ, Kaufman JS, Marshall SW, Gaynes BN, Morrissey JP, Engel CC. Deployment and the use of mental health services among U.S. Army wives. N Engl J Med. 2010 Jan 14;362(2):101-9. doi: 10.1056/NEJMoa0900177. PMID 20071699